CLINICAL TRIAL: NCT03571971
Title: Load Modification Versus Standard Exercise to Inform Treatment for Individuals With Greater Trochanteric Pain Syndrome
Brief Title: Load Modification Versus Standard Exercise for Greater Trochanteric Pain Syndrome
Acronym: GLAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Foundation for Physical Therapy Research (Other)
Responsible Party: Principal Investigator, Stephanie Di Stasi, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017H0450
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Hip Injuries; Pain; Therapy/Rehabilitation
MeSH Terms: conditions — Hip Injuries; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Load modification education (Experimental): Load modification education includes exercises currently prescribed by physical therapists, like stretching and strengthening activities, but will also include education on common daily postures and movement patterns that may increase load and stress on the muscles and tendons around the hip.
  Interventions: Other: Load modification education
- Standard exercise education (Active Comparator): Standard exercise education includes exercises currently prescribed by physical therapists, like stretching and strengthening activities.
  Interventions: Other: Standard exercise education

INTERVENTIONS:
Other: Load modification education — Load modification education includes exercises currently prescribed by physical therapists, like stretching and strengthening activities, but will also include education on common daily postures and movement patterns that may increase load and stress on the muscles and tendons around the hip.
  Other Names: Load modification
  Arms: Load modification education
Other: Standard exercise education — Standard exercise education includes exercises currently prescribed by physical therapists, like stretching and strengthening activities.
  Other Names: Standard exercise
  Arms: Standard exercise education

SUMMARY:
Greater trochanteric pain syndrome (GTPS), or lateral hip pain, is associated with muscle weakness, altered movement patterns and painful daily activities. The disability associated with GTPS is comparable to end stage hip osteoarthritis, primarily affecting young and middle aged women. Few non-operative treatments have demonstrated long-term lasting or satisfactory results. For those who do improve, recurrence rates of pain and disability can be as high as 50%.

Gluteal tendinopathy is the most common condition associated with a GTPS diagnosis. High compressive loads of the gluteal tendons during common activities like walking, stair-climbing, and running are the theorized mechanism for GTPS. These compressive loads are exacerbated with postures and movement patterns that involve the lateral tilting of the pelvis or movement of the thigh across the midline of the body. There is recent evidence that load modification through education and exercise is superior to a corticosteroid injection for reducing pain in these patients. However, it is unknown whether the possible effects of the load modification program were due to exercise alone or the reduction in compressive loads. As current physical therapy interventions for GTPS commonly incorporate high load postures and exercise activities, there is an urgent need to compare outcomes of standard of care physical therapy to load modification.

The goal of this study is to evaluate the short-term effects of load modification education on pain and function in individuals with GTPS. Participants will be randomized to receive either standard exercise education or load modification education. Both groups will complete a series of questionnaires about their pain and function, and undergo a brief 2-dimensional assessment of their posture and movement. Between follow-up sessions, participants will be asked to respond to brief weekly online surveys to document their home program compliance, pain, and function. It is hypothesized that the group of participants receiving load modification will have the highest proportion of individuals with significant improvements in pain and function, and will demonstrate improved posture and movement.

ELIGIBILITY:
Inclusion Criteria: Unilateral diagnosis of GTPS, as confirmed by physician using the following criteria:

* Lateral hip pain, worst over greater trochanter, for >/= 3 months
* Pain with palpation over greater trochanter
* Average pain intensity of >/= 4/10 most days of the week
* Lateral hip pain reproduced during a 30 second single leg stance, or at least one of the following positive tests:

  1. >/= 2/10 lateral hip pain reproduce with passive hip flexion, adduction, and external rotation (ie. FADER)
  2. lateral hip pain reproduced with resisted internal rotation in the passive hip flexion, adduction, and external rotation position (ie. FADER-R)
  3. lateral hip pain reproduce with overpressure into passive hip adduction in sidelying (ie. ADD)
  4. lateral hip pain reproduced with resisted hip abduction in the hip hip adducted position (ie. ADD-R)
  5. lateral hip pain reproduced with hip flexion, abduction, external rotation (ie. FABER)

     Exclusion Criteria:

  <!-- -->

  1. Any of the following treatments within the last 3 months:

     1. corticosteroid injection in the affected hip
     2. physical therapy or other skilled exercise intervention by a medical or rehabilitation professional
  2. Any of the following concomitant impairments or conditions:

     a) Known or observed advanced spine, hip, knee, or ankle joint pathology, including: i. Spinal or lower extremity surgery within the last 6 months ii. Imaging data showing Kellgren Lawrence grade >/=2 in any lower extremity joint with concurrent complaint >/=2/10 most days of the week.

     iii. Groin pain as the primary hip pain complaint >/=2/10 most days of the week.

     iv. <90 degrees of active hip and knee flexion bilaterally v. <0 degrees of active ankle dorsiflexion

     b) Systemic inflammatory diseases, or any systemic disease that affects the nervous or musculoskeletal system or uncontrolled diabetes, or active malignancy c) Individuals who cannot tolerate or should not assume the positions required for the exercises for any reason other than hip discomfort

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Di Stasi, PhD, PT, Principal Investigator — Ohio State University
Locations (1):
- Jameson Crane Sports Medicine Institute, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time, individual participant data (IPD) will be shared only with researchers listed on the funding associated with this project and the Institutional Review Board list of approved key personnel. Deidentified IPD will be made available upon request for purposes of manuscript review and submission. Deidentified IPD may be made available to individuals upon request.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One individual was enrolled and then withdrawn by the study team prior to randomization because they had a systemic condition that met study exclusion criteria. Part of our eligibility assessment process was to consent individuals prior to asking additional questions about their hip problem and other health conditions. We called this our 'step-step' eligibility verification process, and those participants who disclosed information that excluded them from study participation were withdrawn.
Period: Overall Study
Arm/Group | Load Modification Education | Standard Exercise Education
Started | 31 | 30
Completed | 23 | 25
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Incomplete primary outcome data | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Load Modification Education | Standard Exercise Education | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Median (Full Range); unit: years] | 54.4 [27.9 to 69.4] | 57.0 [21.1 to 70.7] | 55.9 [21.1 to 70.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 30 | 27 | 57
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 25 | 23 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 30 | 61
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (9.2) | 30.1 (7.2) | 29.7 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Global Rating of Change
Description: Participant perception of functional change, measured on an 11-point likert scale from 'very much worse' (minimum, worse outcome) to 'very much better' (maximum, better outcome). Results were then dichotomized into those who indicated they were at least 'moderately better' and those who did not.
Time Frame: 4 weeks after enrollment
Population: All participants with Global Rating of Change data at 4 weeks, who also had Numeric Pain Rating Scale data at baseline and 4-weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Load Modification Education | Standard Exercise Education
Number analyzed (Participants) | 23 | 25
Participants
  At least 'moderately better' | 7 | 3
  Were not at least 'moderately better' | 16 | 21
  Did not complete the question | 0 | 1
Statistical Analysis 1: Comparison: Load Modification Education vs Standard Exercise Education; Test type: Superiority — Based on published data, we conservatively estimated that the standard exercise (SE) group and load modification (LM) group would have a 20% and 50% treatment success rate, respectively. We defined treatment success as either: 1) at least 'moderately better' on the Global Rating of Change scale or 2) ≥2 point decrease on the Numeric Pain Rating Scale. With one-side type I error=0.1, power=80%, and allocation ratio is 1:1, we estimated the need for 22 participants in each group (total N=44); p = 0.879, Chi-squared — The a priori threshold for statistical significance was set at 0.05; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.36 to 3.35]

2. Primary Outcome: Change in Numeric Pain Rating Scale
Description: The Numeric Pain Rating Scale (NPRS) is a self-report survey of a participant's worst hip pain in the last week on an 11-point (0-10) scale, where 0 is no pain, 10 is the worst pain imaginable. The Change in NPRS is calculated by subtracting the baseline NPRS from the 4-week NPRS. A positive response to treatment was defined less than or equal to -2 (i.e., pain reduction by 2 points).
Time Frame: at the time of enrollment and 4 weeks after enrollment
Population: We included individuals who had baseline and 4-week Numeric Pain Rating Scale data, and 4-week Global Rating of Change data.
Measure: Count of Participants; unit: Participants
Arm/Group | Load Modification Education | Standard Exercise Education
Number analyzed (Participants) | 23 | 25
Participants
  reported at least 2 point decrease in pain | 10 | 10
  did not report at least 2 point decrease in pain | 13 | 15

3. Secondary Outcome: Change in Pain Self-Efficacy Questionnaire (PSEQ)
Description: The Pain Self-Efficacy Questionnaire is a 10-question survey about confidence with activities of daily living, and each question uses a 7-point likert scale, where 0 represents "not at all confident" and 6 represents "completely confident." Answers to each of the 10 questions are summed to generate a total score. Higher scores represent a better outcome; the best score is 60, the worst score is 0. We used the change in PSEQ from the time of enrollment to 4 weeks after enrollment.
Time Frame: at the time of enrollment and 4 weeks after enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Load Modification Education | Standard Exercise Education
Number analyzed (Participants) | 20 | 24
score on a scale | 3.6 (10.4) | 3.3 (11.1)

4. Secondary Outcome: Change in Victorian Institute of Sport Assessment for Greater Trochanteric Pain Syndrome (VISA-G)
Description: The Victorian Institute of Sport Assessment for Greater Trochanteric Pain Syndrome is a 8-question survey about perceived hip pain and associated functional limitations during various daily activities. Question 1 asks respondents about their usual hip pain severity, scored from 0-10 (1-unit intervals), with 0 represent the worst pain. Questions 2-7 have 5 options that are scored 0, 2, 5, 7, or 10 points, with 0's representing extreme difficulty or inability and 10's representing no difficulty with the activity. Question 8 requires respondents to choose one subsection (A, B, or C) that best corresponds with how their hip pain affects their exercise; the minimum score is 0, the maximum is 30. To calculate the total score, scores from each question are summed. Higher total scores represent a better outcome; the best score is 100, the worst score is 0. We used the change in VISA-G from the time of enrollment to 4 weeks after enrollment.
Time Frame: at the time of enrollment and 4 weeks after enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Load Modification Education | Standard Exercise Education
Number analyzed (Participants) | 21 | 24
score on a scale | 7.7 (13.1) | 1.1 (11.9)

5. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Bank v2.0 Physical Function
Description: The Patient Reported Outcomes Measurement Information System Bank v2.0 Physical Function assesses self-reported physical function of respondents using computerized adaptive testing techniques. It uses responses to each item to calculate a T-score and it is recommended that scoring occur in REDCapTM or similar scoring service to calculate scores using response pattern scoring. The mean score for adults in the United States is 50 with a standard deviation of 10. Higher T-scores are associated with better function and lower T-scores are associated with worse physical function, and T-scores generally range from 20-80. We used the change in PROMIS-PF from the time of enrollment to 4 weeks after enrollment.
Time Frame: at the time of enrollment and 4 weeks after enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Load Modification Education | Standard Exercise Education
Number analyzed (Participants) | 21 | 25
score on a scale | 1.02 (4.04) | 0.73 (4.89)

6. Secondary Outcome: Tegner Activity Level Scale
Description: Tegner Activity Level Scale is a self-report scale of physical activity. The scale has 11 categorical options ranging from complete disability/inactivity (0) to national elite-level sports (11). The best score is 11, indicating elite-level activity participation.
Time Frame: 4 weeks after enrollment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Load Modification Education | Standard Exercise Education
Number analyzed (Participants) | 21 | 24
score on a scale | 3 [3 to 5] | 3 [3 to 5]

7. Secondary Outcome: Patient Acceptable Symptomatic State Question
Description: The Patient Acceptable Symptomatic State is a single question (yes/no response) asking respondents whether or not they are satisfied with their current state, considering all daily activities, their level of pain, and perceived functional impairment. Selecting 'Yes' would indicate the respondent is satisfied with their current state, selecting 'No' would indicate the respondent is not satisfied with their current state.
Time Frame: 4 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Load Modification Education | Standard Exercise Education
Number analyzed (Participants) | 22 | 25
Participants
  Number indicating 'satisified' | 8 | 6
  Number indicating 'not satisfied' | 14 | 19

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 4-week active intervention period during which time the participant received the exercise education (standard or load modification) and engaged in the 4-week home exercise program.
Description: We used adverse event and/or serious adverse event definitions as defined by clinicaltrials.gov. Additionally, we defined an 'Other (Not Including Serious) Adverse Event as either (1) acute onset, severe joint pain or sustain an acute injury during their participation in testing or physical therapy intervention or (2) two consecutive weeks where a participant reported either "moderately worse," "much worse,"or "very much worse" on their weekly Global Rating of Change question.
Arm/Group | Load Modification Education | Standard Exercise Education
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 1/23 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Load Modification Education (N=23) | Standard Exercise Education (N=25)
Musculoskeletal adverse event (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — 1 participant met the following criteria: two consecutive weeks where a participant reports "moderately worse," "much worse," or "very much worse" on their weekly Global Rating of Change question.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT03571971/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT03571971/ICF_001.pdf